CLINICAL TRIAL: NCT01597869
Title: Safety of Endobronchial Ultrasound-guided Transbronchial Needle Aspiration : A Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kyung Jong Lee, professor, Samsung Medical Center
Other Study IDs: 2012-02-009
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Ultrasound; Complication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Endobronchial ultrasound — EBUS-TBNA is a bronchoscopic diagnostic method that enables real time aspiration of paratracheal and peribronchial lesions.

SUMMARY:
The purpose of this study is to find all kinds of complications and it's frequency related to the Endobronchial Ultrasound- Transbronchial Needle Aspiration (EBUS-TBNA) and to evaluate associated risk factors in patients who developed complications. The investigators performs EBUS-TBNA examination on all subjects that need mediastinal evaluation. All complications during or after the procedure will be recorded prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Mediastinal lymph node enlargement on chest CT or PET-CT

Exclusion Criteria:

* Inadequate oxygenation during procedure
* uncontrolled cardiac arrythmia
* Bleeding diathesis
* Severe thrombocytopenia
* Recent use of clopidogrel
* Uncooperative patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admmitted to the tertiary hospital
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Complications related with EBUS-TBNA | 1 month interval
  1. Complications during procedure
     * Bleeding
     * pneumothorax
     * shock
     * cardiac arrythmia
     * change of oxygen saturation
  2. Complication after procedure
     * fever
     * bleeding
     * pneumothorax
     * all other comlications after 24hr

SECONDARY OUTCOMES:
Risk factors related with the development of complications | 1 month interval
  1. Midazolam/Lidocaine dosage
  2. Procedure time
  3. Total aspiration number
  4. Location of sampled lymph node
  5. Sampling number of lymph nodes
  6. Underlying disease
  7. Pulmonary function test

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Jong Lee, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea